CLINICAL TRIAL: NCT07001904
Title: Interleukin-6 in Plaque Psoriasis and Its Possible Role in Disease Severity
Status: Completed | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Adel Jamal Khaled Jadallah, Resident of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Other Study IDs: 36264MS308/9/23
Record Dates: First submitted 2025-05-24; First posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Interleukin-6; Plaque Psoriasis; Disease Severity
MeSH Terms: interventions — Enzyme-Linked Immunosorbent Assay

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients group: Patients with plaque psoriasis.
  Interventions: Other: Enzyme-linked immunosorbent assay (ELISA)
- Control group: Sex- and age-matched healthy control individuals.
  Interventions: Other: Enzyme-linked immunosorbent assay (ELISA)

INTERVENTIONS:
Other: Enzyme-linked immunosorbent assay (ELISA) — The enzyme-linked immunosorbent assay (ELISA) was utilized in order to determine the levels of IL-6 in the serum

SUMMARY:
This study aimed to evaluate serum IL-6 levels in plaque psoriasis patients and investigate their correlation with disease severity.

DETAILED DESCRIPTION:
Psoriasis is a chronic, immune-mediated inflammatory dermatological condition that impacts around 0.2% to 4.8% of the worldwide population.

Interleukin (IL)-6 is a pleiotropic cytokine that regulates immunity, hematopoiesis, and inflammation. It is produced by keratinocytes, endothelial cells, fibroblasts, and immune cells like macrophages and dendritic cells. Increased IL-6 expression has been observed in psoriatic lesions, suggesting its involvement in disease pathogenesis

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years.
* Both sexes.
* Patients clinically diagnosed with plaque psoriasis.

Exclusion Criteria:

* Patients who had received any treatment for psoriasis in the last three months.
* Patients with other types of psoriasis.
* Those currently receiving systemic treatment.
* Individuals with other inflammatory diseases.
* Pregnant or lactating women.
* Those using contraceptive pills.
* Patients with metabolic conditions like diabetes mellitus or thyroid disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This cross-sectional work had been performed on 30 individuals with plaque psoriasis and 20 sex- and age-matched healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Disease severity | 3 months post-procedure
  Disease severity was assessed using the Psoriasis Area and Severity Index (PASI), categorizing patients into mild (PASI <5), moderate (PASI 5-10), and severe (PASI >10) groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.